CLINICAL TRIAL: NCT03328247
Title: Achieving Self-directed Integrated Cancer Aftercare (ASICA) in Melanoma: A Randomized Patient-focused Trial of Delivering the ASICA Intervention as a Means to Earlier Detection of Recurrent and Second Primary Melanoma
Brief Title: Achieving Self-directed Integrated Cancer Aftercare (ASICA) in Melanoma
Acronym: ASICA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aberdeen (Other)
Collaborators: Cancer Research UK (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2-028-17
Record Dates: First submitted 2017-10-23; First posted 2017-11-01 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Control group will attend their routine melanoma follow-ups
- Intervention (Experimental): The intervention group will use the ASICA app in addition to their routine follow-ups
  Interventions: Other: ASICA digital app

INTERVENTIONS:
Other: ASICA digital app — Participants in the intervention arm will be trained to use ASICA (in addition to completing routine follow-up) and participants within the control arm will continue to attend their usual structured melanoma follow-up only. The hypothesis is that the ASICA intervention will increase TSSE practice in those affected by melanoma without affecting psychological well-being and lead to earlier detection of recurrent and new primary melanoma.
  Arms: Intervention

SUMMARY:
The ASICA study is looking at how the UK National Health Service (NHS) might use technology in the future to more effectively support people who have been treated for melanoma.

DETAILED DESCRIPTION:
All patients who have been treated for melanoma are advised to regularly examine their own skin (total-skin-self-examinations; TSSE) but research has found that many people are not shown how to do this effectively. We are investigating whether a digital app we have developed (ASICA) can help people with melanoma to use a hand-held tablet computer to do more regular and effective TSSE, and whether this would lead to earlier detection of recurrent and new primary melanomas. The ASICA app also uses the internet to enable people to electronically communicate the findings of their TSSE to a specialist nurse. All those who consent to take part in the study will be randomly allocated into one of two groups. One group will use the ASICA app in addition to their normal follow-up, the other group will continue to attend their routine melanoma follow-up only. Participants will be recruited from two UK sites - NHS Grampian and Cambridge University Hospitals.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥18)
* Patients treated for stage 0-2C cutaneous melanoma within the preceding 24 months

Exclusion Criteria:

* Stage 3 and 4 melanoma.
* Previous local recurrence of melanoma within last 24 months.
* Patients who are unable to consent and/or complete questionnaires (e.g. due to cognitive or language issues).
* Patients who are blind or visually impaired.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2018-01-12 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
The impact of receiving ASICA on cancer worry | Up to 12 months following randomisation.
  This outcome will be measured using Melanoma Worry Scale (MWS). The scale consists of four questions asking the patients how worried they are about getting melanoma and how this impacts their current lifestyle. The patients choose the answers on a 5-point scale ranging from 'not at all worried' (best answer) to 'worried almost all the time' (worst answer).
The impact of receiving ASICA on anxiety and depression | Up to 12 months following randomisation.
  This outcome will be measured using Hospital Anxiety and Depression Scale (HADS). HADS was devised to measure anxiety and depression in a general medical population of patients. The questionnaire comprises seven questions for anxiety and seven questions for depression. The patients choose the answers on a 4-point scale ranging from 'not at all' (best answer) to 'all the time' (worst answer). Each item on the questionnaire is scored from 0-3 leading to a score range of 0 and 21 for each subscales (anxiety or depression). For both scales, scores of less than 7 indicate non-cases, scores of 8-10 indicate mild anxiety/depression, scores of 11-14 indicate moderate anxiety/depression, and scores of 15-21 indicate severe anxiety/depression.
The impact of receiving ASICA quality of life. | Up to 12 months following randomisation.
  This outcome will be measured using EQ-5D-5L questionnaire. EQ-5D-5L consists of two sections - descriptive system and a visual scale. The descriptive system comprises of five questions about mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each question has five possible answers ranging from: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient chooses the most appropriate statement in each of the five questions. This decision results in a 1-digit number that expresses the level selected for that question. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state. The higher the number the worse the health state is. The visual scale records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The worst health you can imagine' (score of 0) and 'The best health you can imagine' (score of 100).

SECONDARY OUTCOMES:
The impact of receiving ASICA on detection rate of second primary and recurrent melanoma | Up to 12 months following randomisation.
  The questionnaire consists of 14 questions asking patients whether they have ever and in the past 12 month checked any part of their skin for signs of skin cancer (yes/no answer). If so, how often (5 point scale ranging from 'zero' to 'more than six times') and which areas of the body were checked. The patients are also asked whether they used a mirror or get help to check difficult to reach areas of their body. The patients are also asked how confident they are about being able to check their own skin. Patients choose the answers on a 10-point scale ranging from 'not at all confident' (worst answer) to 'highly confident' (best answer). The final set of questions ask patients whether they have found anything concerning during their last skin check (yes/no answer) and if so what action was taken by the patient (watched it/showed it to a relative/showed it to a professional) and how quickly (immediately, in few days, in a week, in a month, other).
The impact of receiving ASICA on adherence to and self-efficacy to conduct TSSE in future | Up to 12 months following randomisation.
  This outcome will be measured using a questionnaire designed to determine what the patients think about examining their own skin. The questionnaire consists of nine statements about how important it is to patients to check their skin, do they do it regularly, does it make them anxious, whether they feel confident about having their skin checked by a professional, and do they make plans regarding when and where they will have their skin checked. For each statement, patients indicate whether they strongly disagree, disagree, agree, strongly agree, or are unsure.
The impact of receiving ASICA on patterns of UK NHS resource use | Up to 12 months following randomisation.
  This outcome will be measured using a questionnaire designed to determine whether patients used NHS because of their skin problems. The set of seven questions is about any appointments within the NHS that patients may have had about their skin in the past 12 months. Patients are asked whether they had any appointments with a medical professional (GP/nurse/other) for their skin in the past 12 months (yes/no answer), how many (free text) and at what setting (visit at the practice/visit at home/telephone). Patients are also asked about operations or any other treatment they may have had on their skin in the past 12 months (free text). Patients are also asked to list any prescribed medicines or non-prescribed skin products in the last 12 months and their cost (free text).

CONTACTS AND LOCATIONS:
Overall Officials: Peter Murchie, MBChB, PhD, Principal Investigator — University of Aberdeen
Locations (2):
- United Kingdom (2):
  - University of Aberdeen, Aberdeen
  - Addenbrookes Hospital, Cambridge

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Reilly F, Wani N, Hall S, Morgan HM, Allan J, Constable L, Ntessalen M, Murchie P. User Experiences in a Digital Intervention to Support Total Skin Self-examination by Melanoma Survivors: Nested Qualitative Evaluation Embedded in a Randomized Controlled Trial. JMIR Dermatol. 2023 Feb 13;6:e39544. doi: 10.2196/39544. PMID 37632942
- [Derived] Ntessalen M, McCorkindale S, Krasniqi A, Morgan HM, Allan JL, Murchie P. Barriers and facilitators of adherence to the use of ASICA, a digital app designed to support people previously treated for melanoma: concise report of a qualitative study. Clin Exp Dermatol. 2023 Nov 16;48(12):1358-1360. doi: 10.1093/ced/llad279. PMID 37611174
- [Derived] Murchie P, Constable L, Hall S, Brant W, Allan J, Johnston M, Masthoff J, Lee A, Treweek S, Ayansina D, Proby C, Rahman K, Walter F, Burrows N, Durrani A, Maclennan G. The Achieving Self-directed Integrated Cancer Aftercare Intervention for Detection of Recurrent and Second Primary Melanoma in Survivors of Melanoma: Pilot Randomized Controlled Trial. JMIR Cancer. 2022 Sep 8;8(3):e37539. doi: 10.2196/37539. PMID 36074560
- [Derived] Allan JL, Johnston DW, Johnston M, Murchie P. Describing, predicting and explaining adherence to total skin self-examination (TSSE) in people with melanoma: a 12-month longitudinal study. BMJ Open. 2022 Aug 30;12(8):e056755. doi: 10.1136/bmjopen-2021-056755. PMID 36041758
- [Derived] Reilly F, Contstable L, Brant W, Rahman K, Durrani A, Burrows N, Proby C, Allan J, Johnston M, Johnston D, Walter F, Murchie P. Achieving integrated self-directed Cancer aftercare (ASICA) for melanoma: how a digital intervention to support total skin self-examination was used by people treated for cutaneous melanoma. BMC Cancer. 2021 Nov 13;21(1):1217. doi: 10.1186/s12885-021-08959-2. PMID 34774015
- [Derived] Murchie P, Masthoff J, Walter FM, Rahman K, Allan JL, Burrows N, Proby C, Lee AJ, Johnston M, Durrani A, Depasquale I, Brant B, Neilson A, Meredith F, Treweek S, Hall S, McDonald A. Achieving Self-Directed Integrated Cancer Aftercare (ASICA) in melanoma: protocol for a randomised patient-focused pilot trial of delivering the ASICA intervention as a means to earlier detection of recurrent and second primary melanoma. Trials. 2019 Jun 3;20(1):318. doi: 10.1186/s13063-019-3453-x. PMID 31159849